CLINICAL TRIAL: NCT03894761
Title: What Are the Factors Affecting Night Pain in Patients With Rotator Cuff Syndrome
Brief Title: Night Pain in Patients With Rotator Cuff Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Alper Mengi, Medical Doctor, Physiatrist, Gaziosmanpasa Research and Education Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13.06.18/69
Record Dates: First submitted 2019-03-21; First posted 2019-03-29 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Shoulder Pain; Shoulder Impingement Syndrome; Shoulder Tendinitis; Rotator Cuff Tear
Keywords: Pain; Shoulder; Rotator Cuff
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome; Rotator Cuff Injuries; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Rotator Cuff Syndrome (Other): The patients diagnosed with rotator cuff syndrome by clinical and magnetic resonance imaging.
  Interventions: Other: Night Pain in Patients with Rotator Cuff Syndrome

INTERVENTIONS:
Other: Night Pain in Patients with Rotator Cuff Syndrome — The pain severity was evaluated using a 10 cm visual analogue scale , where 0 represented no pain, while 10 represented unbearable pain.At evaluation, the average of the pain during night for the last one week were inquired.

SUMMARY:
The aim of this study is to determine the factors that may be associated with night pain in patients diagnosed with rotator cuff syndrome by clinical and magnetic resonance imaging.

DETAILED DESCRIPTION:
Patients who were diagnosed as rotator cuff syndrome by clinical examination and magnetic resonance imaging will be included in this prospective study.

Demographic data (gender, age, education level, occupation), shoulder pain duration, history of trauma to the shoulder, smoking, dominant arm and diabetes will be questioned and body mass indexes will be calculated. Active shoulder range of motion of the patients will be measured by goniometer and recorded .

Specific tests, which are important for rotator cuff lesion, will be performed to determine whether they are positive or not.

Magnetic resonance imaging of the patients with shoulder pathology will be recorded.

A visual analog scale will be used to determine the intensity of day and night pain. Shoulder Shoulder Pain and Disability Index to assess shoulder disability of patients, SF-36 form will be filled by patient to evaluate the effect of shoulder pathology and Kinesiophobia Score to assess the avoidance of pain induced movement.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with rototor cuff pathology by magnetic resonance imaging
* Age range between 18-65 years old
* To be literate and cooperative

Exclusion Criteria:

* Having shoulder pathology other than rototor cuff pathology (Glenohumeral instability, Bisipital tendon lesions, Glenohumeral joint osteoarthritis, Acromioclavicular joint osteoarthritis, Milwaukee shoulder)
* Having complete rotator cuff tear
* Patients with a history of shoulder or cervical surgery
* The presence of cervical pathology
* Patients with a history of fracture in the shoulder with pain
* Local corticosteroid injection history for the shoulder (over the last 6 months) and using painkiller regularly
* Physical therapy history for the shoulder (in the last 3 months)
* The presence of systemic inflammatory disease
* Malignancy
* Pregnancy
* A history of any psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Night pain: visual analogue scale | 7 day
  The pain severity was evaluated using a 10 cm visual analogue scale , where 0 represented no pain, while 10 represented unbearable pain.At evaluation, the average of the pain during night for the last one week were inquired.

SECONDARY OUTCOMES:
Demographic datas | 1 day
  Gender, Age, Education Level, Job
Daytime pain: visual analogue scale | 7 day
  The pain severity was evaluated using a 10 cm visual analogue scale , where 0 represented no pain, while 10 represented unbearable pain.At evaluation, the average of the pain during daytime for the last one week were inquired.
Range of Motion of the Shoulder | 1 day
  The shoulder range of motion of the patients will be measured in the form of active range of motion and using a goniometer. The shoulder range of motion will be measured as flexion, extension, internal rotation, external rotation, abduction and adduction.
Pathology in magnetic resonance imaging | 1 day
  The rotator cuff pathologies will be evaluated in MR imaging as subacromial-subdeltoid effusion, supraspinatus muscle tendinosis, supraspinatus muscle tear, supraspinatus muscle calcific tendinitis, infraspinatus muscle tendinosis, infraspinatus muscle tear, teres minör muscle tendinosis, teres minör muscle tear, subscapularis muscle tendinosis, subscapularis muscle tear.
The Shoulder Pain and Disability Index | 7 days
  The Shoulder Pain and Disability Index (SPDA) is a self-administered questionnaire that consists of two dimensions (for pain and for functional activities). The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use.
  Each of the 13 items is to be rated with a number from 0 to 10:
  * For the pain score (first 5 items): 0 means no pain and 10 means worst pain imaginable;
  * For the disability score (last 8 items): 0 means no impairment and 10 means the patient requires help to perform that action.
  Scores could theoretically range from 0 to 100 with higher scores indicating greater impairment. The total SPADI score was calculated by averaging the pain and disability subscale scores. The total SPADI score could also range from 0 to 100.
Tampa Scale of Kinesiophobia | 7 days
  Tampa Scale of Kinesiophobia is a 17-item self report checklist using a 4-point Likert scale that was developed as a measure of fear of movement or (re)injury.
  The TSK is a self-completed questionnaire and the range of scores are from 17 to 68 where the higher scores indicate an increasing degree of kinesiophobia.
The Short Form-36 | 7 days
  Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Body mass index | 1 day
  The formula is Body mass index = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.
pain duration | 1 day
  The duration of pain will be asked to patients as months.
history of trauma to the shoulder | 1 day
  It will be questioned whether patients had a history of trauma to the shoulder before.
dominant hand and affected arm side | 1 day
  The patients will be asked which hands are dominant (right or left), and the side with shoulder pain (right or lelft) will be recorded.
smoking history | 6 months
  Patients will be asked about their smoking habit for the last 6 months.
diabetes history | 1 day
  The patients will be asked whether they have diabetes disease.
Hawkins test | 1 day
  Hawkins test is performed by elevating the patient's arm forward to 90 degrees while forcibly internally rotating the shoulder. Patients will be evaluated for positive test or negative test.
Neer test | 1 day
  Neer test is performed by placing the arm in forced flexion with the arm fully pronated . The scapula is stabilized during the maneuver to prevent scapulothoracic motion. Patients will be evaluated for positive test or negative test.
Painful arc test | 1 day
  The patient fully abducts their arm in the scapular plane , and is considered positive if the patient reports pain between 60 degrees and 120 degrees of abduction.
Jobe test | 1 day
  The patient's arm elevates to 90 degrees in the scapular plane, with the elbow extended, full internal rotation, and pronation of the forearm. This results in a thumbs-down position, as if the patient were pouring liquid out of a can, and the patient tries to resist this motion. This test is considered positive if the patient experiences pain or weakness with resistance.
drop-arm test | 1 day
  This test is performed by passively abducting the patient's shoulder, then observing as the patient slowly lowers the arm to the waist. Patients will be evaluated for positive test or negative test.
Patte test | 1 day
  The examiner places the patient's arm to 90 degrees in the scapular plane and flexes the elbow to 90 degrees . The patient is then asked to externally rotate against resistance. The test is positive if the patient is unable to perform external rotation.
External rotation test | 1 day
  The examiner passively flexes the patient's elbow to 90 degrees and brings the shoulder into a position of 20 degrees of scaption. Next, the examiner passively takes the patient's shoulder into a position of maximal lateral rotation. The patient in then instructed to hold that position. A positive test is if the patient cannot maintain the position and the shoulder rotates internally.
Lag sign test | 1 day
  The elbow is passively flexed to 90° and the shoulder abducted to 90° and held 5° off maximal external rotation. The patient is then asked to maintain the position actively while the examiner releases the wrist while maintaining support through the elbow.Patients will be evaluated for positive test or negative test.
Gerber lift-off test | 1 day
  The patient is examined in standing and is asked to place their hand behind their back with the dorsum of the hand resting in the region of the mid- lumbar spine. The dorsum of the hand is raised off the back by maintaining or increasing internal rotation of the humerus and extension at the shoulder.
  Inability to move the dorsum off the back constitutes an abnormal lift-off test and indicates subscapularis rupture or dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Mengi, M.D., Principal Investigator — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Alper Mengi, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No